CLINICAL TRIAL: NCT00967889
Title: Molecular Mechanisms of Disease Progression and the Development of Novel Treatment Strategies in Advanced Prostate Cancer (Northern Prostate Cancer Collaborative (ProMPT))
Brief Title: Study of Tissue, Blood, and Urine Samples From Patients With Advanced Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CRUK-ProMPT; CDR0000638974 (Registry Identifier: PDQ (Physician Data Query)); EU-20919
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Prostate Cancer
Keywords: stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gene Expression Profiling

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: protein analysis
Other: biologic sample preservation procedure
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue, blood, and urine from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat the cancer.

PURPOSE: This research study is looking at tissue, blood, and urine samples from patients with advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To study molecular pathology and mechanisms of disease progression.
* To develop novel treatment strategies for patients with advanced prostate cancer.
* To evaluate novel markers and treatment and epidemiological approaches.

OUTLINE: This is a multicenter study.

* Program I (Molecular Signaling in Advanced Prostate Cancer): Researchers from Newcastle, York, and Bristol analyze androgen receptor (AR) (i.e., AR regulated genes and AR co-activators and co-repressors) and fibroblast growth factor (FGF) signaling and examine the cross-talk between these two systems and the insulin-like growth factor (IGF) axis.
* Program II (Mechanisms of Skeletal Metastases): Researchers from Newcastle, Sheffield, Bristol, and Manchester analyze mechanisms of skeletal metastases and candidate factors responsible for skeletal metastases (e.g., BMP-6, TGF-β1, IL-6, and IL-6 receptor). The balance between proteases and their inhibitors is also analyzed.
* Program III (Prostate Targeting, Models, and Novel Approaches to Therapy): Researchers from Newcastle, Sheffield, York, and Manchester analyze and develop reagents and methods that will facilitate novel gene-based approaches to therapy, including prostate tissue specific gene expression, model systems of gene function and therapeutic studies, translational gene-based therapies, and effectors for potential gene therapy.
* Program IV (Developmental Therapeutics): Researchers from Newcastle, York, and Manchester analyze novel proteins identified during the study to synthesize novel reagents aimed at disrupting pathways and signaling molecules that have been shown to be of critical importance to prostate cancer (e.g., AR and FGF signaling).
* Program V (Biorepository and Database): Tissue, DNA, blood, serum, and urine samples from Newcastle, Sheffield, and Manchester biorepositories are stored and used for analysis in programs I-IV. Support for tissue and data collection as well as database management is provided to enable these resources to be made available to the wider research community.
* Program VI (Clinical Trials and Health Services Research): Researchers from Newcastle, Sheffield, Manchester, and Bristol participate in phase I trials using dendritic cells and gene-directed enzyme prodrug therapy (GDEPT) approaches to analyze environmental interactions with the genotype and evaluate prevention strategies (e.g., diet) that may underlie variations in the incidence of prostate cancer.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced prostate cancer

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-01; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Molecular pathology and mechanisms of disease progression
Development of novel treatment strategies for patients with advanced prostate cancer
Evaluation of novel markers and treatment and epidemiological approaches

CONTACTS AND LOCATIONS:
Overall Officials: David Neil, MD, Principal Investigator — Cancer Research UK
Locations (1):
- Cancer Research UK at Cambridge Research Institute, Cambridge, England, United Kingdom